CLINICAL TRIAL: NCT06848075
Title: A Phase IIb, Randomized, Double-Blind, Placebo-Controlled Study of Elismetrep (K-304) in the Treatment of Migraine: A Range of Doses Will be Evaluated
Brief Title: A Phase IIb, Randomized, Double-Blind, Placebo-Controlled Study of Elismetrep (K-304) in the Treatment of Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kallyope Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K-304 P001
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Acute Migraine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Elismetrep (K-304) Dose level 1 (Experimental)
  Interventions: Drug: Elismetrep (K-304) Dose Level 1
- Elismetrep (K-304) Dose level 2 (Experimental)
  Interventions: Drug: Elismetrep (K-304) Dose level 2
- Elismetrep (K-304) Dose level 3 (Experimental)
  Interventions: Drug: Elismetrep (K-304) Dose level 3
- Elismetrep (K-304) Dose level 4 (Experimental)
  Interventions: Drug: Elismetrep (K-304) Dose level 4
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Elismetrep (K-304) Dose Level 1 — Administered orally
  Arms: Elismetrep (K-304) Dose level 1
Drug: Elismetrep (K-304) Dose level 2 — Administered orally
  Arms: Elismetrep (K-304) Dose level 2
Drug: Elismetrep (K-304) Dose level 3 — Administered orally
  Arms: Elismetrep (K-304) Dose level 3
Drug: Elismetrep (K-304) Dose level 4 — Administered orally
  Arms: Elismetrep (K-304) Dose level 4
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, multicenter, outpatient evaluation of the safety and efficacy of elismetrep as compared to placebo in the treatment of moderate or severe migraine.

ELIGIBILITY:
Inclusion Criteria:

1. Be a male or female, age 18 to 70 years, inclusive, at the time of signing informed consent.
2. Patient has greater than a one-year history of migraine with or without aura as defined by International Conference on Harmonization (IHS) criteria 1.1 and 1.2 and his/her migraines typically last between 4 to 72 hours, if untreated as documented in the patient's medical records from his/her treating physician and confirmed by the investigator.
3. Patient has had ≥2 and ≤10 moderate or severe migraine attacks per month in each of the two months prior to screening (Visit 1).
4. Meet the following requirements:

   1. Is a male OR
   2. Is a female who is of non-childbearing potential defined by at least 1 of the following criteria:
   3. Postmenopausal (aged >45 years and with a minimum of 12 months of spontaneous amenorrhea with a Screening serum follicle-stimulating hormone (FSH) level in the menopausal range established for the central laboratory.
   4. Post hysterectomy, bilateral oophorectomy or bilateral salpingectomy, based on the subject's recall of their medical history.

      OR
   5. Is a female of reproductive potential and:
   6. agrees to remain abstinent from heterosexual activity*

      *Abstinence can be used as the sole method of contraception if it is in line with the subject's preferred and usual lifestyle and if considered acceptable by local regulatory agencies and ethics committees. Periodic abstinence (e.g., calendar, ovulation, sympto-thermal, post-ovulation methods, etc.) and withdrawal are not acceptable methods of contraception.
   7. or agrees to use (or have their partner use) a birth control method that is acceptable from the first dose of study drug until the end of trial (EoT) visit. Acceptable methods of birth control are:

      * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

        * oral
        * intravaginal
        * transdermal
      * progestogen-only hormonal contraception associated with inhibition of ovulation:

        * oral
        * injectable
        * implantable
      * intrauterine device (IUD)
      * intrauterine hormone-releasing system (IUS)
      * bilateral tubal occlusion
      * vasectomised partner
      * sexual abstinence
      * progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action
      * male or female condom with or without spermicide
      * cap, diaphragm or sponge with spermicide
      * A combination of male condom with either cap, diaphragm or sponge with spermicide (double barrier methods)

   This condition is waived if the subject is proven to have no child-bearing potential (eg, hysterectomy).
5. Patient voluntarily agrees to participate in the study by giving written informed consent.
6. Patient is able to read, understand and complete the study questionnaires and diary.
7. Be willing and able to comply with the study schedule of visits, all trial procedures and restrictions.
8. Be willing to use their own personal, qualified smartphone to download study specific eDiary applications for use during the study.

Exclusion Criteria:

1. Is a female who is pregnant, breast-feeding or intends to become pregnant during the planned course of the study. Note: Participants must have a negative serum pregnancy test (β-human chorionic gonadotropin (β-hCG)) performed by the central laboratory prior to enrollment in the study and negative urine pregnancy result at the randomization visit.

   Migraine history-related
2. Patient has difficulty distinguishing his/her migraine attacks from tension-type headaches.
3. Patient has a history of predominantly mild migraine attacks or migraines that usually resolve spontaneously in less than two hours.
4. Patient has more than 15 headache-days per month or has taken medication for acute headache on more than 10 days per month in any of the three months prior to screening (Visit 1).
5. Patient has brainstem (a.k.a. basilar-type) or hemiplegic migraine headache, or retinal migraine.
6. Patient was >50 years old at age of first migraine onset.
7. Patient is taking migraine prophylactic medication where the prescribed daily dose has changed during the 3 months prior to screening (Visit 1) or anticipates any change during the study. Any withdrawal of preventive medications for the treatment of migraine should be completed at least 30 days prior to screening.

   Medical history related
8. Patient has, in the opinion of the investigator, other confounding pain syndromes, psychiatric conditions such as uncontrolled major depression, history of psychosis, dementia or significant neurological disorders other than migraine. [Patients who are currently being treated with non-prohibited medication for depression and symptoms are well controlled, in the opinion of the investigator, are eligible to participate in this study].
9. Patient is at imminent risk of self-harm, based on clinical interview and responses on the Columbia Suicidality Severity Rating Scale (C-SSRS), or of harm to others in the opinion of the investigator. Patients must be excluded if they report suicidal ideation with intent, with or without a plan (i.e., Type 4 or 5 on the C-SSRS) in the past 2 months or suicidal behavior in the past 6 months.
10. Has a recent history (within the past 3 years of the screening visit) or current diagnosis or evidence of endocrine, hematological, immunological, renal, respiratory, neurologic, gastrointestinal, biliary, or genitourinary abnormalities or diseases that, per the investigator's judgement, may jeopardize the subject's safety or compliance with the protocol, or otherwise interfere with interpretation of efficacy and/or safety results.
11. Has a history of malignant neoplasms within the past 5 years prior to screening. Basal and squamous cell skin cancer and any carcinoma in-situ are allowed if they have received treatment and follow-up consistent with local standard of care.
12. Patient history with current evidence of uncontrolled, unstable or recently diagnosed cardiovascular disease, such as ischemic heart disease, coronary artery vasospasm, and cerebral ischemia. Patients with Myocardial Infarction (MI), Acute Coronary Syndrome (ACS), percutaneous Coronary Intervention (PCI), cardiac surgery, stroke or transient ischemic attack (TIA) during the 6 months prior to screening.
13. Has a history of human immunodeficiency virus disease.
14. Patient has a history of gastric or small intestinal surgery (including gastric bypass surgery or banding but not including cholecystectomy or appendectomy) or has a disease that causes malabsorption.

    Laboratory, vital sign, and electrocardiogram (ECG) related
15. Has a positive test result at Screening for hepatitis B surface antigen (Ag), hepatitis C virus antibody.
16. Has a screening estimated Glomerular Filtration Rate (eGFR) estimated with the Modification of Diet in Renal Disease (MDRD) equation of <45 ml/min/1.73 m2.
17. Has a screening result for alanine aminotransferase or aspartate aminotransferase (ALT or AST) of >2.0X upper limit of normal (ULN) or total bilirubin >1.5X ULN at the Screening visit. Note: An isolated bilirubin >1.5X ULN is acceptable if bilirubin is fractionated, and direct bilirubin is within the laboratory normal range.
18. Has a corrected QT interval to Fridericia's formula (QTcF) >450 milliseconds (msec) for males and >470 msec for females at screening.
19. Has a mean value for triplicate seated systolic blood pressure >160 mmHg and/or diastolic blood pressure (BP) >95 mmHg measured after at least 5 minutes at rest at the Screening Visit.

    Note: If a subject's BP is exclusionary on the first triplicate assessment at the Screening visit, they may have 1 repeat triplicate BP assessment at that visit after another rest of at least 10 minutes.

    Medication use and substance abuse related
20. Has known history of or suspected abuse of alcohol or recreational drugs at Screening.
21. Has use of soft drugs (such as marijuana or any substances containing tetrahydrocannabinol (THC) or cannabidiol (CBD)) within 3 months prior to Screening, or hard drugs (such as cocaine, illicit narcotics/opiates) within 6 months prior to Screening.
22. Has a positive drug screen at Screening. Note: If benzodiazepines are detected on the drug screen, this is not exclusionary if they are prescribed a benzodiazepine for a therapeutic purpose (e.g. for insomnia) and confirmatory documentation is obtained from the prescribing physician.
23. Is currently in violation of study requirements for prohibited and permissible concomitant medications (not already specified in other criteria) or is anticipated to violate these requirements during study participation.
24. Has any use of prescription opiate medications within 14 days of screening or any anticipated/potential use of opiates during study participation.
25. History of use of ergotamine medications on greater than/equal 10 days per month on a regular basis for greater than/equal 3 months prior to screening.
26. History of non-narcotic analgesic intake on greater than/equal 15 days per month for greater than/equal 3 months prior to screening.

    Other
27. Has known or suspected hypersensitivity to trial product(s) or related products.
28. Has a history of multiple significant and/or any severe allergies (e.g., food, drug, latex allergy) or has had an anaphylactic reaction or significant intolerance to prescription or nonprescription drugs or food.
29. Has any surgery scheduled for the duration of the trial.
30. Had major surgery or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the Screening Visit; has a screening hemoglobin <11.0 g/dL (males) or <10.0 g/dL (females), or has a known hemoglobinopathy (e.g. sickle cell anemia, hemolytic anemia).
31. Has previous participation in this trial. Participation is defined as signed informed consent.
32. Has participated in any clinical trial of an approved or non-approved investigational biological medicinal product (e.g. antibody therapy) within 90 days of Screening or has participated in any clinical trial of an approved or non-approved investigational small molecule medicinal product within 30 days or 5 half-lives (whichever is longer) of Screening.
33. Has any other disorder, unwillingness or inability, not covered by any of the other exclusion criteria, which in the investigator's opinion, might jeopardize the subject's safety or compliance with the protocol, or otherwise interfere with interpretation of efficacy and/or safety results.
34. Is an employee or immediate family member (e.g., spouse, parent, child, sibling) of the Sponsor or study site.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Pain freedom | 2 hours post-dose
  Assessed using the number of evaluable subjects that report no pain

SECONDARY OUTCOMES:
Freedom from the most bothersome symptom (MBS) (nausea, phonophobia or photophobia) | 2 hours post-dose
  Assessed using the number of evaluable subjects that report the absence of their MBS
Pain relief | 2 hours post-dose
  Assessed using the number of evaluable subjects that report a pain level of moderate or severe (responses of 2 or 3 on the 4-point Likert scale) at baseline and then report a pain level of none or mild (response of 0 or 1)
Freedom from Photophobia | 2 hours post-dose
  Assessed by tabulating the number of subjects that report the absence of photophobia at 2 hours post-dose in the subset of subjects that reported the presence of photophobia at headache baseline
Freedom from Phonophobia | 2 hours post-dose
  Assessed by tabulating the number of subjects that report the absence of phonophobia at 2 hours post-dose in the subset of subjects that reported the presence of phonophobia at headache baseline
Freedom from Nausea | 2 hours post-dose
  Assessed by tabulating the number of subjects that report the absence of nausea at 2 hours post-dose in the subset of subjects that reported the presence of nausea at headache baseline
The probability of requiring rescue medication | 24 hours post-dose
  Assessed using the number of subjects that take rescue medication within 24 hours after administration of study medication
Sustained pain freedom | From 2 to 24 hours
  Assessed using the number of subjects that do not experience any headache pain through the time period of interest
Sustained pain relief | From 2 to 24 hours
  Assessed using the number of subjects that do not experience any moderate or severe headache pain through the time period of interest
Sustained pain freedom | From 2 to 48 hours
  Assessed using the number of subjects that do not experience any headache pain through the time period of interest
Sustained pain relief | From 2 to 48 hours
  Assessed using the number of subjects that do not experience any moderate or severe headache pain through the time period of interest
Proportion of participants who experienced 1 or more treatment-emergent AEs | up to 7 days after administration of study medication
Proportion of participants who experienced 1 or more treatment-emergent SAEs | up to 7 days after administration of study medication

CONTACTS AND LOCATIONS:
Locations (66):
- United States (66):
  - Central Research Associates, LLC (CRA) dba Flourish Research, Birmingham, Alabama
  - AMR Mobile, Mobile, Alabama
  - Wake Research/ Tucson Neuroscience Research, Tucson, Arizona
  - Hope Clinical Research, Canoga Park, California
  - WR-PRI, LLC (Encino), Encino, California
  - Marvel Clinical Research, Huntington Beach, California
  - Eximia Research - CA, La Mesa, California
  - Synergy San Diego, Lemon Grove, California
  - WR-PRI, LLC (Newport Beach), Newport Beach, California
  - Excell Research, Inc., Oceanside, California
  - Empire Clinical Research, Pomona, California
  - Artemis Institute for Clinical Research - Riverside, Riverside, California
  - Acclaim Clinical Research, San Diego, California
  - Artemis Institute for Clinical Research - San Diego, San Diego, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Focus Clinical Research, West Hills, California
  - CT Clinical Research, Cromwell, Connecticut
  - DelRicht Research, Atlanta, Georgia
  - Clinical Research Atlanta - Stockbridge, Stockbridge, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Cedar Crosse Research Center, Chicago, Illinois
  - Healthcare Research Network II, LLC, Flossmoor, Illinois
  - Collective Medical Research, Overland Park, Kansas
  - Alliance for Multispecialty Research, Wichita, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Crescent City Headache & Neurology Center, Chalmette, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Michigan Head Pain and Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - DelRicht Research, Gulfport, Mississippi
  - Healthcare Research Network, Hazelwood, Missouri
  - Excel Clinical Research, Las Vegas, Nevada
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Dent Neurosciences Research Center, Amherst, New York
  - CNY Clinical Research, Manlius, New York
  - Rochester Clinical Research, Rochester, New York
  - Upstate Clinical Research Associates LLC, Williamsville, New York
  - Headache Wellness Center, Greensboro, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - OK Clinical Research, LLC, Edmond, Oklahoma
  - Hightower Clinical, Oklahoma City, Oklahoma
  - DelRicht Research, Tulsa, Oklahoma
  - Tekton Research, Yukon, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Clinical Research Philadelphia, LLC, Philadelphia, Pennsylvania
  - Frontier Clinical Research, LLC, Scottdale, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Atlas-Clinical, West Chester, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - WR-ClinSearch, Chattanooga, Tennessee
  - AMR Knoxville (Formerly NOCCR), Knoxville, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Donald J Garcia Jr, MD, PA, Austin, Texas
  - Tekton Research, Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Victorium Clinical Research LTD CO, Houston, Texas
  - APD Clinical Research, Splendora, Texas
  - ClinPoint Trials, Waxahachie, Texas
  - Advanced Research Institute, Ogden, Utah
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Frontier Clinical Research, LLC, Morgantown, West Virginia
  - Clinical Investigation Specialist, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No